CLINICAL TRIAL: NCT01634828
Title: Method for Improved Intraoperative Blood Loss Estimates
Acronym: EBL
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Annette Macintyre, Principle Investigator, University of Utah
Other Study IDs: FP00002762; 56181 (Registry Identifier: IRB University of Utah)
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Improved Intraoperative Blood Loss Estimates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Minimal blood loss patients
- Moderate to heavy blood loss patients

SUMMARY:
The purpose of this study is to develop a mathematical algorithm which the investigators plan to use to more accurately estimate intraoperative blood loss.

ELIGIBILITY:
Inclusion Criteria:

All elective surgical patients

Exclusion Criteria:

1. Age < 18
2. Pregnant women
3. Prisoners
4. Lack of informed consent
5. Attending Physician feels enrollment could interfere with optimal patient care
6. Patients who did not have a preoperative hemoglobin measured as part of their preoperative work-up
7. Patients whose preoperative hemoglobin fraction is abnormal.
8. Patients who will likely require an intraoperative blood transfusion.
9. Patients for whom the intraoperative use of the Cell Saver is anticipated.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elective surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Estimate of intraoperative blood loss | duration of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States